CLINICAL TRIAL: NCT00005936
Title: Collection of Liver Tissue for Virologic Studies
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000167; 00-H-0167
Record Dates: First submitted 2000-07-06; First posted 2000-07-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-03

CONDITIONS: Virus Disease
Keywords: Fulminant Hepatitis; Parvovirus; Hepatitis; Biopsy; Control; Liver Biopsy
MeSH Terms: conditions — Virus Diseases; Massive Hepatic Necrosis; Parvoviridae Infections; Hepatitis

SUMMARY:
This study will examine liver tissue to investigate the role of viral infections in fulminant hepatitis, liver failure, and profound bone marrow failure.

All patients who are undergoing liver biopsy or liver transplantation may participate in this study. For patients undergoing liver biopsy, a small piece of liver tissue will be taken from the sample collected during the scheduled biopsy. For patients undergoing liver transplantation, a small piece of tissue will be collected from the diseased liver that is to be removed.

DETAILED DESCRIPTION:
Our laboratory has a long-standing interest in viruses that affect the bone marrow. Many such viruses also may cause hepatitis. One specific syndrome, post-hepatitis aplastic anemia, suggests that the same agent is responsible for both severe and sometimes fulminant hepatitis as well as profound bone marrow failure. In investigating the role of viruses in these diseases, we require small amounts of liver tissue for molecular studies. We request permission to obtain samples from patients undergoing 1) liver transplantation or 2) liver biopsy at the time of surgery for purpose of virus discovery, including obtaining control samples. For liver transplant samples, tissue will be obtained from the removed organ; in other surgical circumstances, small amounts of tissue will be obtained when the liver is biopsied for other medical indications. No additional risk to the patient should result from either procedure.

ELIGIBILITY:
All patients undergoing open liver biopsy or the removal of liver for purposes of hepatic transplantation are eligible for participation.

There are no exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2000-06; Study Completion 2002-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Naides SJ, Karetnyi YV, Cooling LL, Mark RS, Langnas AN. Human parvovirus B19 infection and hepatitis. Lancet. 1996 Jun 1;347(9014):1563-4. doi: 10.1016/s0140-6736(96)90720-5. No abstract available. PMID 8684141
- [Background] Tzakis AG, Arditi M, Whitington PF, Yanaga K, Esquivel C, Andrews WA, Makowka L, Malatak J, Freese DK, Stock PG, et al. Aplastic anemia complicating orthotopic liver transplantation for non-A, non-B hepatitis. N Engl J Med. 1988 Aug 18;319(7):393-6. doi: 10.1056/NEJM198808183190702. PMID 3135496
- [Background] Brown KE, Tisdale J, Barrett AJ, Dunbar CE, Young NS. Hepatitis-associated aplastic anemia. N Engl J Med. 1997 Apr 10;336(15):1059-64. doi: 10.1056/NEJM199704103361504. PMID 9091802